CLINICAL TRIAL: NCT00630422
Title: Functional Abilities in Rett Syndrome
Status: Completed | Type: Observational
Sponsor: Faculdades Metropolitanas Unidas (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: carlos bandeira de mello monteiro, Faculdades Metropolitanas Unidas
Other Study IDs: monteiro; monteiro1
Record Dates: First submitted 2008-01-17; First posted 2008-03-07 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-01

CONDITIONS: Rett Syndrome
Keywords: Rett Syndrome; Selfcare; Mobility limitation; Interpersonal relations; This study avaliated patients with Rett Syndrome
MeSH Terms: conditions — Rett Syndrome; Mobility Limitation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 64: All Patients

SUMMARY:
The purpose of this study is to evaluate and determinate the functional abilities in Rett syndrome conforming to the established Pediatric Evaluation of Disability Inventory (PEDI).

DETAILED DESCRIPTION:
Rett syndrome (RS) is a progressive neurological disturbance of genetic cause that affects females almost exclusively. It is caused by mutations, usually sporadic, of the MECP2 gene located in the X chromosome. In consequence to the serious cognitive and motor compromise, the RS patients have great difficulty in accomplishing day-to-day tasks. The objective of this work is to evaluate the functional abilities in RS to help therapists in theirs treatments programs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Rett syndrome that matched the criteria for the classic form of the disease

Exclusion Criteria:

* Any other disease;
* Rett syndrome associated with other disease
* Rett syndrome that not that matched the criteria for the classic form of the disease

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study investigated only patients with Rett syndrome that matched the criteria for the classic form of the disease
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2006-02; Primary Completion 2006-09 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, PhD, Principal Investigator — Faculdades Metropolitanas Unidas
Locations (1):
- Faculdades Metropolitanas Unidas, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: alread published — http://www.teses.usp.br/teses/disponiveis/5/5138/tde-28052007-150911/